CLINICAL TRIAL: NCT06256016
Title: Application of Massage to the Dorsal Paravertebral Muscles and Its Efficacy in the Treatment of Neck Pain
Brief Title: Effectiveness of Massage of the Thoracic Region in Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Prof. Dr. Daniel Pecos Martín, Principal investigator, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEI15/002
Record Dates: First submitted 2024-02-04; First posted 2024-02-13 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neck pain massage (Experimental): Subjects in this group will be treated with a neck muscle massage protocol.
  Interventions: Other: Neck pain massage
- Neck and thoracic massage (Experimental): Subjects in this group will be treated with a massage protocol of the neck muscles and the posterior thoracic region.
  Interventions: Other: Neck and thoracic massage

INTERVENTIONS:
Other: Neck pain massage — Subjects in this group will be treated with a neck muscle massage protocol. First, pressure inhibition techniques will be applied to the affected muscles. Then deep stroke technique will be performed on each muscle.
  In addition, effleurages technique will be applied along the thoracic paravertebral muscle.
  Subjects will also perform an exercise protocol for neck pain.
  Arms: Neck pain massage
Other: Neck and thoracic massage — Subjects in this group will be treated with a neck muscle massage protocol. First, pressure inhibition techniques will be applied to the affected muscles. Then deep stroke technique will be performed on each muscle.
  In addition, deep stroke technique will be applied along the thoracic paravertebral muscle.
  Subjects will also perform an exercise protocol for neck pain.
  Arms: Neck and thoracic massage

SUMMARY:
Neck pain is a common disorder in industrialized countries. Manual therapy techniques have been commonly used in the treatment of this problem. Actually, there is no research work that has evaluated the work well of treatment with soft tissue techniques (massage) applied to the dorsal paravertebral muscle in the management of neck pain. The goal of this study (clinical trial) is to compare the efficacy of a massage protocol performed on the dorsal region in subjects with mechanical neck pain.

The researchers will compare:

A group that will be treated with a local protocol of cervical manual therapy and therapeutic exercise along with the treatment(massage) of the thoracic region.

Another group that will be treated only with a local protocol of cervical manual therapy and therapeutic exercise.

It is to see if the inclusion of treatment of the thoracic region improves the local intervention in cervical region.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with neck pain.
* Pain between 4 and 7 points according to a visual anological scale.
* Neck pain lasting more than three months

Exclusion Criteria:

* Subjects who have suffered a whiplash injury.
* Subjects with neck pain and upper extremity pain.
* Subjects with a diagnosis of herniated disc.
* Subjects with fibromyalgia.
* Subjects with any cancer process.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Neck pain | Change from Baseline pain at 3 month
  A Visual Analogue Scale (VAS) is one of the pain rating scales used for measure the intensity pain. The VAS is a straight horizontal line of fixed length, usually 100 mm.The ends are defined as the extreme limits of the parameter to be measured orientated from the left or "10" (worst pain) to the right (best pain) or "0".

SECONDARY OUTCOMES:
Neck disability index | Change from Baseline pain at 3 month
  This questionnaire has been designed to give us information as to how the neck pain are affecting the subject´s ability to manage in everyday life. The questionnaire has 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. It´s interpreted as a raw score, with a maximum score of 50 where "0" is not disability and 50 is the worst disability
Pain catastrophizing | Change from Baseline pain at 3 month
  Pain Catastrophizing Scale (PCS). The PCS is a 13-item instrumen that task participants to reflect on past painful experiences, and to indicate the degree to which they experienced each of 13 thoughts or feelings when experiencing pain, on 5-point scales with the end points (0) not at all and (4) all the time. The PCS total scores range from 0 - 52. 0 is the best result and 52 is the worst result.
kinesiophobia | Change from Baseline pain at 3 month
  The Tampa Scale of Kinesiophobia (TSK) describe patient circumstances characterised by an "excessive, irrational, and debilitating fear of physical movement and activity resulting from a feeling of vulnerability to painful injury or reinjury. The TSK is a 17 item assessment checklist.The 17 item TSK total scores range from 17 to 68 where the lowest 17 means no or negligible kinesiophobia, and the higher scores indicate an increasing degree of kinesiophobia.
The Global Rating of Change (GRoC) | Change from Baseline pain at 3 month
  It's a scale that assesses whether the patient condition has gotten worse, better, or stayed the same and to quantify the magnitude of that change, typically following treatment.Subjects will make global ratings of changes regarding their level of well-being from their neck pain since the initial examination on a 15-point self-report scale (from -7 to 7), where -7 is the worst possible value and 7 is the best possible value.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Pecos-Martin, PhD, Principal Investigator — Alcala University
Locations (1):
- Physioterapy and Pain center research, Alcalá de Henares, Madrid, Spain